CLINICAL TRIAL: NCT06430801
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled Program to Evaluate the Efficacy and Safety of Tulisokibart in Participants With Moderately to Severely Active Crohn's Disease
Brief Title: A Study to Evaluate the Efficacy and Safety of Tulisokibart (MK-7240) in Participants With Moderate to Severe Crohn's Disease (MK-7240-008)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 7240-008; MK-7240-008 (Other: MSD); 2023-508636-61-00 (Registry Identifier: EU CT); U1111-1298-6080 (Registry Identifier: UTN); jRCT2031240196 (Registry Identifier: jRCT)
Record Dates: First submitted 2024-05-21; First posted 2024-05-28 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Crohn's Disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (11):
- Study 1: High Dose Induction, High Dose Maintenance (Experimental): Participants receive high dose intravenous (IV) tulisokibart, followed by a high dose subcutaneous (SC) tulisokibart regimen.
  Interventions: Drug: IV Tulisokibart; Drug: SC Tulisokibart
- Study 1: High Dose Induction, Low Dose Maintenance (Experimental): Participants receive high dose IV tulisokibart, followed by a low dose SC tulisokibart regimen.
  Interventions: Drug: IV Tulisokibart; Drug: SC Tulisokibart; Other: SC Placebo
- Study 1: Low Dose Induction, Low Dose Maintenance (Experimental): Participants receive low dose IV tulisokibart, followed by a low dose SC tulisokibart regimen.
  Interventions: Drug: IV Tulisokibart; Drug: SC Tulisokibart; Other: SC Placebo
- Study 1: Placebo (Placebo Comparator): Participants receive IV placebo, followed by an SC placebo regimen.
  Interventions: Drug: IV Tulisokibart; Other: IV Placebo; Other: SC Placebo
- Study 1: High Dose Extension (Experimental): Participants receive a high dose SC tulisokibart regimen. Participants may continue in this arm after completing participation in their original arm, if they meet protocol-specific prerequisites.
  Interventions: Drug: SC Tulisokibart
- Study 1: Low Dose Extension (Experimental): Participants receive a low dose SC tulisokibart and placebo regimen. Participants may continue in this arm after completing participation in their original arm, if they meet protocol-specific prerequisites.
  Interventions: Drug: SC Tulisokibart; Other: SC Placebo
- Study 2: High Dose Induction (Experimental): Participants receive high dose IV tulisokibart.
  Interventions: Drug: IV Tulisokibart
- Study 2: Low Dose Induction (Experimental): Participants receive low dose IV tulisokibart.
  Interventions: Drug: IV Tulisokibart; Other: SC Placebo
- Study 2: Placebo (Placebo Comparator): Participants receive IV placebo.
  Interventions: Drug: IV Tulisokibart; Other: IV Placebo; Other: SC Placebo
- Study 2: High Dose Extension (Experimental): Participants receive a high dose SC tulisokibart regimen. Participants may continue in this arm only after completing participation in their original arm, if they meet protocol-specific prerequisites.
  Interventions: Drug: SC Tulisokibart
- Study 2: Low Dose Extension (Experimental): Participants receive a low dose SC tulisokibart regimen. Participants may continue in this arm only after completing participation in their original arm, if they meet protocol-specific prerequisites.
  Interventions: Drug: SC Tulisokibart

INTERVENTIONS:
Drug: IV Tulisokibart — Humanized monoclonal antibody that binds human tumor necrosis factor-like cytokine 1A (TL1A), administered intravenously
  Other Names: PRA023; MK-7240
  Arms: Study 1: High Dose Induction, High Dose Maintenance; Study 1: High Dose Induction, Low Dose Maintenance; Study 1: Low Dose Induction, Low Dose Maintenance; Study 1: Placebo; Study 2: High Dose Induction; Study 2: Low Dose Induction; Study 2: Placebo
Drug: SC Tulisokibart — Humanized monoclonal antibody that binds human TL1A, administered subcutaneously
  Other Names: PRA023; MK-7240
  Arms: Study 1: High Dose Extension; Study 1: High Dose Induction, High Dose Maintenance; Study 1: High Dose Induction, Low Dose Maintenance; Study 1: Low Dose Extension; Study 1: Low Dose Induction, Low Dose Maintenance; Study 2: High Dose Extension; Study 2: Low Dose Extension
Other: IV Placebo — Placebo matching IV tulisokibart
  Arms: Study 1: Placebo; Study 2: Placebo
Other: SC Placebo — Placebo matching SC tulisokibart
  Arms: Study 1: High Dose Induction, Low Dose Maintenance; Study 1: Low Dose Extension; Study 1: Low Dose Induction, Low Dose Maintenance; Study 1: Placebo; Study 2: Low Dose Induction; Study 2: Placebo

SUMMARY:
The purpose of this protocol is to evaluate the efficacy and safety of tulisokibart in participants with moderately to severely active Crohn's disease. Study 1's primary hypotheses are that at least 1 tulisokibart dose level is superior to placebo in the proportion of participants achieving clinical remission per Crohn's Disease Activity Index score (<150, US/FDA) or per stool frequency and abdominal pain score (EU/EMA) and in the proportion of participants achieving endoscopic response at Week 52 (US/FDA and EU/EMA), and that at least 1 tulisokibart dose level is superior to placebo in the proportion of participants achieving clinical remission per Crohn's Disease Activity Index score (<150, US/FDA) or per stool frequency and abdominal pain score (EU/EMA) and in the proportion of participants achieving endoscopic response at Week 12 (US/FDA and EU/EMA). Study 2's primary hypothesis is that at least 1 tulisokibart dose level is superior to placebo in the proportion of participants achieving clinical remission per Crohn's Disease Activity Index score (<150, US/FDA) or stool frequency and abdominal pain score (EU/EMA) and in the proportion of participants achieving endoscopic response at Week 12 (US/FDA and EU/EMA).

DETAILED DESCRIPTION:
The protocol consists of 2 studies. Study 1 includes induction and maintenance treatment, and Study 2 includes only induction treatment. Each study has its own hypotheses and outcome measures that will be assessed independently.

ELIGIBILITY:
The main inclusion and exclusion criteria include but are not limited to the following:

Inclusion Criteria:

* Has had a diagnosis of CD at least 3 months before study.
* Has moderately to severely active CD.
* Demonstrated inadequate response, loss of response, or intolerance to one or more of the following categories of drugs: oral locally acting steroids, systemic steroids, immunomodulators, biologic and/or small molecule advanced therapies.
* Adolescent participants ≥16 and <18 years of age can participate if approved by the country or regulatory/health authority.

Exclusion Criteria:

* Has diagnosis of ulcerative colitis (UC) or indeterminate colitis.
* Has CD isolated to the stomach, duodenum, jejunum, or perianal region, without colonic and/or ileal involvement.
* Currently has any of the following complications of CD: suspected or diagnosed with intra-abdominal or perianal abscess, known symptomatic stricture or colonic stenosis not passable in endoscopy, fulminant colitis, toxic megacolon, or any other manifestation that might require surgery while enrolled in the study.
* Has current stoma or need for colostomy or ileostomy.
* Is missing >2 segments of the following 5 segments: terminal ileum, right colon, transverse colon, sigmoid and left colon, and rectum.
* Has been diagnosed with short gut or short bowel syndrome, or any other uncontrolled chronic diarrhea besides Crohn's disease.
* Has surgical bowel resection within 3 months of study.
* Has prior or current gastrointestinal dysplasia.
* Has chronic infection requiring ongoing antimicrobial treatment.
* Has a history of cancer (except fully treated non-melanoma skin cell cancers or cervical carcinoma in situ after complete surgical removal) and is disease free for <5 years.
* Is infected with Hepatitis B virus (HBV), Hepatitis C virus (HCV), or human immunodeficiency virus (HIV).
* Has active tuberculosis.
* Has confirmed or suspected coronavirus disease of 2019 (COVID-19) infection.
* Prior exposure to tulisokibart (MK-7240, PRA023) or another anti-TL1A antibody.

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2024-06-05 (Actual); Primary Completion 2028-10-30 (Estimated); Study Completion 2029-11-12 (Estimated)

PRIMARY OUTCOMES:
Study 1 [US/FDA Only]: Percentage of Participants Achieving Clinical Remission per Crohn's Disease Activity Index (CDAI) Score at Week 52 | Week 52
  The percentage of participants achieving clinical remission, as defined by CDAI score <150 for study 1 will be presented.
Study 1 [EU/EMA Only]: Percentage of Participants Achieving Clinical Remission per Stool Frequency and Abdominal Pain Score at Week 52 | Week 52
  The percentage of participants achieving clinical remission per stool frequency/abdominal pain score (SF/APS), as defined by average daily SF ≤2.8 and average daily APS ≤1.0 and both not greater than baseline for study 1 will be presented.
Study 1: Percentage of Participants Achieving Endoscopic Response at Week 52 | Week 52
  The percentage of participants achieving endoscopic response, as defined by a ≥50% decrease in Simplified endoscopic score for Crohn's disease (SES-CD) from baseline for study 1 will be presented.
Study 1: Percentage of Participants Achieving Clinical Remission per CDAI Score at Week 12 | Week 12
  The percentage of participants achieving clinical remission, as defined by CDAI score <150 for study 1 will be presented.
Study 1: Percentage of Participants Achieving Clinical Remission per Stool Frequency and Abdominal Pain Score at Week 12 | Week 12
  The percentage of participants achieving clinical remission per SF/APS, as defined by average daily SF ≤2.8 and average daily APS ≤1.0 and both not greater than baseline for study 1 will be presented.
Study 1: Percentage of Participants Achieving Endoscopic Response at Week 12 | Week 12
  The percentage of participants achieving endoscopic response, as defined by a ≥50% decrease in SES-CD from baseline for study 1 will be presented.
Study 2 [US/FDA Only]: Percentage of Participants Achieving Clinical Remission per CDAI Score at Week 12 | Week 12
  The percentage of participants achieving clinical remission, as defined by CDAI score <150 for study 2 will be presented.
Study 2 [EU/EMA Only]: Percentage of Participants Achieving Clinical Remission per Stool Frequency and Abdominal Pain Score at Week 12 | Week 12
  The percentage of participants achieving clinical remission per SF/APS, as defined by average daily SF ≤2.8 and average daily APS ≤1.0 and both not greater than baseline for study 2 will be presented.
Study 2: Percentage of Participants Achieving Endoscopic Response at Week 12 | Week 12
  The percentage of participants achieving endoscopic response, as defined by a ≥50% decrease in SES-CD from baseline for study 2 will be presented.

SECONDARY OUTCOMES:
Study 1: Percentage of Participants Who Experienced an Adverse Event (AE) | Up to approximately 52 weeks
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention. The percentage of participants who experience an AE for study 1 will be presented.
Study 1: Percentage of Participants who Discontinue Study Intervention due to an AE | Up to approximately 52 weeks
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention. The percentage of participants who discontinue study intervention due to an AE for study 1 will be presented.
Study 1 [US/FDA Only]: Percentage of Participants Achieving Clinical Remission per Stool Frequency and Abdominal Pain Score at Week 12 | Week 12
  The percentage of participants achieving clinical remission per SF/APS, as defined by average daily SF ≤2.8 and average daily APS ≤1.0 and both not greater than baseline for study 1 will be presented.
Study 1 [EU/EMA Only]: Percentage of Participants Achieving Clinical Remission per CDAI Score at Week 12 | Week 12
  The percentage of participants achieving clinical remission, as defined by CDAI score <150 for study 1 will be presented.
Study 1: Percentage of Participants with Decrease of ≥100 Points in CDAI Score from Baseline to Week 12 | Week 12
  The percentage of participants achieving a reduction in CDAI ≥100 points from baseline for study 1 will be presented.
Study 1: Mean Change from Baseline in Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-Fatigue) Score at Week 12 | Baseline and Week 12
  The FACIT-Fatigue is a 13-item measure that assesses self-reported fatigue and its impact upon daily activities and function, scored on a 0 to 52-point scale, with lower scores indicating greater fatigue. The mean change from baseline in FACIT-Fatigue score for study 1 will be presented.
Study 1: Percentage of Participants Achieving Endoscopic Remission at Week 12 | Week 12
  The percentage of participants achieving endoscopic remission, as defined by SES-CD ≤4 and at least 2-point reduction from baseline and no subscore >1 in any individual variable for study 1 will be presented. SES-CD evaluates 4 endoscopic variables (ulcer size, ulcerated surface, affected surface, and narrowing), each on a scale from 0 to 3, in 5 segments assessed during ileocolonoscopy (ileum, right colon, transverse colon, left colon/sigmoid, and rectum). The total score is the sum of the 4 endoscopic variable scores and ranges from 0 to 56, where higher scores indicate more severe disease.
Study 1 and 2: Percentage of Participants in Diagnostic Assay Positive (Dx+) Subpopulation Achieving Clinical Remission per CDAI at Week 12 | Week 12
  Dx+ participants are those who meet protocol-specific diagnostic assay criteria during screening. The percentage of Dx+ participants achieving clinical remission, as defined by CDAI score <150 for study 1 and study 2 will be presented.
Study 1 and 2: Percentage of Participants in Diagnostic Assay Positive (Dx+) Subpopulation Achieving Endoscopic Response at Week 12 | Week 12
  Dx+ participants are those who meet protocol-specific diagnostic assay criteria during screening. The percentage of Dx+ participants achieving endoscopic response, as defined by a ≥50% decrease in simplified endoscopic score for Crohn's disease (CD) from baseline for study 1 and study 2 will be presented.
Study 1 [US/FDA Only]: Percentage of Participants Achieving Clinical Remission per Stool Frequency and Abdominal Pain Score at Week 52 | Week 52
  The percentage of participants achieving clinical remission per SF/APS, as defined by average daily SF ≤2.8 and average daily APS ≤1.0 and both not greater than baseline for study 1 will be presented.
Study 1: Percentage of Participants Achieving Clinical Remission per CDAI Score at Week 52 | Week 52
  The percentage of participants achieving clinical remission, as defined by CDAI score <150 for study 1 will be presented.
Study 1: Percentage of Participants with Decrease of ≥100 Points in CDAI Score from Baseline to Week 52 | Week 52
  The percentage of participants achieving a reduction in CDAI ≥ 100 points from baseline for study 1 will be presented.
Study 1: Percentage of Participants Achieving Endoscopic Remission at Week 52 | Week 52
  The percentage of participants achieving endoscopic remission, as defined by SES-CD ≤4 and at least 2-point reduction from baseline and no subscore >1 in any individual variable for study 1 will be presented. SES-CD evaluates 4 endoscopic variables (ulcer size, ulcerated surface, affected surface, and narrowing), each on a scale from 0 to 3, in 5 segments assessed during ileocolonoscopy (ileum, right colon, transverse colon, left colon/sigmoid, and rectum). The total score is the sum of the 4 endoscopic variable scores and ranges from 0 to 56, where higher scores indicate more severe disease.
Study 1: Percentage of Participants Achieving Sustained Clinical Remission per CDAI at Both Week 12 and Week 52 | Week 12 and Week 52
  The percentage of participants achieving sustained clinical remission, as defined by CDAI score <150 for study 1 will be presented.
Study 1: Percentage of Participants Achieving Corticosteroid-Free Clinical Remission per CDAI Score at Week 52 | Week 52
  The percentage of participants who are in clinical remission as defined by CDAI score <150 and without corticosteroid use for CD at least 90 days prior to that assessment for study 1 will be presented.
Study 1: Percentage of Participants Achieving Corticosteroid-Free Clinical Remission per Stool Frequency and Abdominal Pain Score at Week 52 | Week 52
  The percentage of participants who are in clinical remission per SF/APS, as defined by average daily SF ≤2.8 and average daily APS ≤1.0 and both not greater than baseline and without corticosteroid use for CD at least 90 days prior to that assessment for study 1 will be presented.
Study 1: Percentage of Participants Achieving Clinical Remission per Stool Frequency, Abdominal Pain Score, and Endoscopic Remission at Week 52 | Week 52
  The percentage of participants achieving clinical remission per SF/APS, as defined by average daily SF ≤2.8 and average daily APS ≤1.0 and both not greater than baseline and achieving endoscopic remission, as defined by SES-CD ≤4 and at least 2-point reduction from baseline and no subscore >1 in any individual variable for study 1 will be presented.
Study 1: Percentage of Participants Achieving Clinical Remission per CDAI and Endoscopic Remission at Week 52 | Week 52
  The percentage of participants achieving clinical remission as defined by CDAI score <150 and achieving endoscopic remission, as defined by SES-CD ≤4 and at least 2-point reduction from baseline and no subscore >1 in any individual variable for study 1 will be presented.
Study 1: Mean Change from Baseline in FACIT-Fatigue Score at Week 52 | Baseline and Week 52
  The FACIT-Fatigue is a 13-item measure that assesses self-reported fatigue and its impact upon daily activities and function, scored on a 0 to 52-point scale, with lower scores indicating greater. The mean change from baseline in FACIT-Fatigue score for study 1 will be presented.
Study 1: Mean Change from Baseline in Inflammatory Bowel Disease Questionnaire (IBDQ) Score at Week 52 | Baseline and Week 52
  The IBDQ measures health related quality of life in participants with inflammatory bowel disease. It consists of 32 questions each with a graded response of 1 (worst) to 7 (best). The score ranges between 32 to 224 with higher scores indicating a better quality of life. The mean change from baseline in IBDQ score for study 1 will be presented.
Study 1: Percentage of Participants with Ulcer-Free Endoscopy at Week 52 | Week 52
  The percentage of participants achieving ulcer-free endoscopy (mucosal healing), as defined by SES-CD ulcerated surface subscore of 0 in participants with SES-CD ulcerated surface subscore ≥1 at baseline for study 1 will be presented.
Study 2: Percentage of Participants Who Experienced an AE | Up to approximately 12 weeks
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention. The percentage of participants who experience an AE for study 2 will be presented.
Study 2: Percentage of Participants who Discontinue Study Intervention due to an AE | Up to approximately 12 weeks
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention. The percentage of participants who discontinue study intervention due to an AE for study 2 will be presented.
Study 2 [US/FDA Only]: Percentage of Participants Achieving Clinical Remission per Stool Frequency and Abdominal Pain Score at Week 12 | Week 12
  The percentage of participants achieving clinical remission per SF/APS, as defined by average daily SF ≤2.8 and average daily APS ≤1.0 and both not greater than baseline for study 2 will be presented.
Study 2 [EU/EMA Only]: Percentage of Participants Achieving Clinical Remission per CDAI Score at Week 12 | Week 12
  The percentage of participants achieving clinical remission, as defined by CDAI score <150 for study 2 will be presented.
Study 2: Percentage of Participants with Decrease of ≥100 Points in CDAI Score from Baseline to Week 12 | Week 12
  The percentage of participants achieving a reduction in CDAI ≥ 100 points from baseline for study 2 will be presented.
Study 2: Mean Change from Baseline in FACIT-Fatigue Score at Week 12 | Baseline and Week 12
  The FACIT-Fatigue is a 13-item measure that assesses self-reported fatigue and its impact upon daily activities and function, scored on a 0 to 52-point scale, with lower scores indicating greater. The mean change from baseline in FACIT-Fatigue score for study 2 will be presented.
Study 2: Percentage of Participants Achieving Endoscopic Remission at Week 12 | Week 12
  The percentage of participants achieving endoscopic remission, as defined by SES-CD ≤4 and at least 2-point reduction from baseline and no subscore >1 in any individual variable for study 2 will be presented. SES-CD evaluates 4 endoscopic variables (ulcer size, ulcerated surface, affected surface, and narrowing), each on a scale from 0 to 3, in 5 segments assessed during ileocolonoscopy (ileum, right colon, transverse colon, left colon/sigmoid, and rectum). The total score is the sum of the 4 endoscopic variable scores and ranges from 0 to 56, where higher scores indicate more severe disease.
Study 2: Mean Change from Baseline in Inflammatory Bowel Disease Questionnaire (IBDQ) Score at Week 12 | Baseline and Week 12
  The IBDQ measures health related quality of life in participants with inflammatory bowel disease. It consists of 32 questions each with a graded response of 1 (worst) to 7 (best). The score ranges between 32 to 224 with higher scores indicating a better quality of life. The mean change from baseline in IBDQ score for study 2 will be presented.
Study 2: Percentage of Participants with Decrease of ≥100 Points in CDAI Score from Baseline to Week 6 | Week 6
  The percentage of participants achieving a reduction in CDAI ≥ 100 points from baseline for study 2 will be presented.
Study 2: The percentage of Participants with Ulcer-Free Endoscopy at Week 12 | Week 12
  The percentage of participants achieving ulcer-free endoscopy (mucosal healing), as defined by SES-CD ulcerated surface subscore of 0 in participants with SES-CD ulcerated surface subscore ≥1 at baseline for study 1 will be presented.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (493):
- United States (81):
  - Digestive Health Specialists ( Site 5064), Dothan, Alabama
  - Arizona Arthritis & Rheumatology Research, PC ( Site 5094), Phoenix, Arizona
  - GI Alliance - Sun City ( Site 5118), Sun City, Arizona
  - University of Arizona Clinical and Translational Sciences Research Center ( Site 5111), Tucson, Arizona
  - Clinnova Research ( Site 5110), Anaheim, California
  - Southern California Research Center ( Site 5044), Coronado, California
  - Om Research LLC ( Site 5038), Lancaster, California
  - Cedars Sinai Medical Center ( Site 5080), Los Angeles, California
  - UCLA Clinical & Translational Research Center (CTRC) ( Site 5116), Los Angeles, California
  - University of California, Irvine (UCI) Health - UC Irvine Medical Center ( Site 5128), Orange, California
  - Om Research LLC ( Site 5045), Oxnard, California
  - Clinical Applications Laboratories ( Site 5123), San Diego, California
  - Amicis Research Center ( Site 5055), Valencia, California
  - University of Colorado Anschutz Medical Campus-Division of Gastroenterology and Hepatology ( Site 5026), Aurora, Colorado
  - Peak Gastroenterology Associates ( Site 5023), Colorado Springs, Colorado
  - South Denver Gastroenterology, PC ( Site 5132), Englewood, Colorado
  - Rocky Mountain Gastroenterology ( Site 5082), Lakewood, Colorado
  - Medical Research Center of Connecticut ( Site 5005), Hamden, Connecticut
  - Yale University School of Medicine-Digestive Disease ( Site 5019), New Haven, Connecticut
  - Emerson Clinical Research Institute ( Site 5051), Washington D.C., District of Columbia
  - Gastroenterology Consultants of Clearwater ( Site 5052), Clearwater, Florida
  - Nature Coast Clinical Research - Inverness ( Site 5042), Inverness, Florida
  - Atlantic Medical Research ( Site 5073), Margate, Florida
  - Sanchez Clinical Research ( Site 5144), Miami, Florida
  - Endoscopic Research Inc ( Site 5061), Orlando, Florida
  - Orlando Health-Digestive Health Institute ( Site 5010), Orlando, Florida
  - USF Health Carol and Frank Morsani Center for Advanced Healthcare ( Site 5039), Tampa, Florida
  - Covenant Metabolic Specialists, LLC ( Site 5143), University Park, Florida
  - Morehouse School Of Medicine ( Site 5071), Atlanta, Georgia
  - Atlanta Center for Gastroenterology ( Site 5035), Decatur, Georgia
  - Gastroenterology Associates of Central Georgia ( Site 5048), Macon, Georgia
  - Eagle Clinical Research ( Site 5089), Chicago, Illinois
  - University of Chicago Medical Center ( Site 5066), Chicago, Illinois
  - Endeavor Health ( Site 5018), Evanston, Illinois
  - GI ALLIANCE - GURNEE ( Site 5003), Gurnee, Illinois
  - Indiana University Health University Hospital ( Site 5022), Indianapolis, Indiana
  - Iowa Digestive Disease Center ( Site 5007), Clive, Iowa
  - University of Kansas Medical Center ( Site 5091), Kansas City, Kansas
  - Cotton O'Neil Digestive Health Center ( Site 5033), Topeka, Kansas
  - University of Louisville Hospital ( Site 5120), Louisville, Kentucky
  - Southern Clinical Research ( Site 5095), Zachary, Louisiana
  - Walter Reed National Military Medical Center ( Site 5006), Bethesda, Maryland
  - Massachusetts General Hospital-Crohn's and Colitis Center ( Site 5037), Boston, Massachusetts
  - University of Michigan ( Site 5060), Ann Arbor, Michigan
  - Clinical Research Institute of Michigan, LLC ( Site 5002), Clinton Township, Michigan
  - Mayo Clinic in Rochester, Minnesota ( Site 5024), Rochester, Minnesota
  - Mid-America GI Clinical Research ( Site 5130), Kansas City, Missouri
  - BVL Research - Kansas ( Site 5099), Liberty, Missouri
  - Washington University School of Medicine ( Site 5058), St Louis, Missouri
  - HMH Justice Marie Garibaldi Medical Plaza ( Site 5072), Hackensack, New Jersey
  - Northwell Health Physician Partners Center for Advanced IBD Care ( Site 5017), Great Neck, New York
  - Circuit Clinical /Crystal Run Healthcare LLP ( Site 5050), Middletown, New York
  - NYU Langone Health - Inflammatory Bowel Disease Center (IBD) ( Site 5078), New York, New York
  - Weill Cornell Medical College, New-York Presbyterian Hospital ( Site 5079), New York, New York
  - New York Gastroenterology Associates ( Site 5013), New York, New York
  - University of North Carolina Medical Center ( Site 5034), Chapel Hill, North Carolina
  - Atrium Health Gastroenterology MMP ( Site 5105), Charlotte, North Carolina
  - Javara - Tryon Medical Partners ( Site 5046), Charlotte, North Carolina
  - Great Lakes Gastroenterology Research, LLC ( Site 5016), Mentor, Ohio
  - Digestive Disease Specialists Inc. ( Site 5117), Oklahoma City, Oklahoma
  - Thomas Jefferson University Hospital ( Site 5133), Philadelphia, Pennsylvania
  - Frontier Clinical Research, LLC ( Site 5098), Uniontown, Pennsylvania
  - University Gastroenterology - Providence - West River Street ( Site 5057), Providence, Rhode Island
  - Sanford USD Medical Center ( Site 5129), Sioux Falls, South Dakota
  - Vanderbilt Inflammatory Bowel Disease Clinic ( Site 5049), Nashville, Tennessee
  - Quality Medical Research ( Site 5114), Nashville, Tennessee
  - Baylor University Medical Center ( Site 5031), Dallas, Texas
  - GI Alliance - Dallas - Gaston Avenue ( Site 5054), Dallas, Texas
  - Baylor College of Medicine Medical Center ( Site 5020), Houston, Texas
  - Michael E. DeBakey VA Medical Center ( Site 5086), Houston, Texas
  - GI Alliance - Lubbock ( Site 5012), Lubbock, Texas
  - Caprock Gastro Research ( Site 5077), Lubbock, Texas
  - GI Alliance: Mansfield ( Site 5015), Mansfield, Texas
  - Southern Star Research Institute ( Site 5000), San Antonio, Texas
  - GI Alliance - Southlake ( Site 5109), Southlake, Texas
  - Tyler Research Institute ( Site 5001), Tyler, Texas
  - Richmond VA Medical Center ( Site 5021), Richmond, Virginia
  - Washington Gastroenterology - Bellevue ( Site 5040), Bellevue, Washington
  - Swedish Medical Center ( Site 5112), Seattle, Washington
  - University of Washington ( Site 5115), Seattle, Washington
  - Washington Gastroenterology - Tacoma ( Site 5004), Tacoma, Washington
- Australia (6):
  - Concord Repatriation General Hospital-Gastroenterology and Liver Services ( Site 3202), Concord, New South Wales
  - Royal Brisbane and Women's Hospital ( Site 3200), Brisbane, Queensland
  - Mater Misericordiae Limited ( Site 3209), Brisbane, Queensland
  - Royal Adelaide Hosp - GI Clinical Trials ( Site 3203), Adelaide, South Australia
  - Monash Health-Gastroenterology ( Site 3206), Clayton, Victoria
  - The Alfred Hospital-Gastroenterology ( Site 3201), Melbourne, Victoria
- Austria (3):
  - Medizinische Universitaet Innsbruck-Innere Medizin 1 ( Site 0200), Innsbruck, Tyrol
  - Medizinische Universität Wien-Klinik für Innere Medizin III - Abteilung für Gastroenterologie und H ( Site 0202), Vienna, Vienna
  - Uniklinikum Salzburg-Innere Medizin I ( Site 0201), Salzburg
- Belgium (3):
  - UZ Gent ( Site 0300), Ghent, Oost-Vlaanderen
  - UZ Leuven-Gastroenterology - Inflammatory Bowel Disease ( Site 0301), Leuven, Vlaams-Brabant
  - AZ Delta vzw-Gastroenterology ( Site 0304), Roeselare, West-Vlaanderen
- Brazil (9):
  - Hospital de Clinicas de Porto Alegre ( Site 6310), Porto Alegre, Rio Grande do Sul
  - Hospital Ernesto Dornelles ( Site 6312), Porto Alegre, Rio Grande do Sul
  - Faculdade de Medicina da UNESP ( Site 6308), Botucatu, São Paulo
  - Loema Instituto de Pesquisa Clinica ( Site 6302), Campinas, São Paulo
  - CECIP - Centro de Estudos do Interior Paulista ( Site 6316), Jaú, São Paulo
  - Hospital das Clínicas da Faculdade de Medicina de Ribeirão Preto da Universidade de São Paulo (USP) ( Site 6311), Ribeirão Preto, São Paulo
  - Pesquisare Saude ( Site 6304), Santo André, São Paulo
  - Centro de Pesquisa Kaiser - CEPEK ( Site 6306), São José do Rio Preto, São Paulo
  - BR Trials - Ensaios Clinicos e Consultoria ( Site 6301), São Paulo
- Canada (17):
  - Heritage Medical Research Clinic ( Site 0004), Calgary, Alberta
  - Gastroenterology and internal medicine research institute ( Site 0009), Edmonton, Alberta
  - Prairie Institute of Liver and Luminal Advanced Research ( Site 0015), Lethbridge, Alberta
  - Fraser Clinical Trials Inc ( Site 0001), New Westminster, British Columbia
  - G.I.R.I. GI Research Institute Foundation ( Site 0018), Vancouver, British Columbia
  - Private Practice - Dr. Bruce Musgrave ( Site 0014), Kentville, Nova Scotia
  - Barrie GI Associates ( Site 0016), Barrie, Ontario
  - University Hospital - London Health Sciences Centre ( Site 0002), London, Ontario
  - London Health Sciences Centre ( Site 0007), London, Ontario
  - West GTA Research Inc. ( Site 0020), Mississauga, Ontario
  - ABP Research Services Corp. ( Site 0019), Oakville, Ontario
  - Toronto Immune & Digestive Health Institute ( Site 0005), Toronto, Ontario
  - Toronto Digestive Disease Associates ( Site 0006), Vaughan, Ontario
  - Centre de recherche du CISSS de Chaudière-Appalaches - Hôpital Hôtel Dieu de Levis ( Site 0011), Lévis, Quebec
  - Centre Hospitalier de l'Université de Montréal - Gastroenterology ( Site 0013), Montreal, Quebec
  - Montreal General Hospital ( Site 0003), Montreal, Quebec
  - Diex Recherche Quebec ( Site 0008), Québec, Quebec
- Chile (8):
  - Clínica Universidad de Los Andes ( Site 2609), Las Condes, Region M. de Santiago
  - FALP-UIDO ( Site 2600), Santiago, Region M. de Santiago
  - Clínica Alemana de Santiago-Unidad de Investigaciones ( Site 2602), Santiago, Region M. de Santiago
  - Espacio Eme ( Site 2608), Santiago, Region M. de Santiago
  - CECIM ( Site 2603), Santiago, Region M. de Santiago
  - Hospital hernan henriquez aravena de temuco ( Site 2607), Temuco, Región de la Araucanía
  - Centro de Investigaciones Clinicas Vina del Mar ( Site 2606), Viña del Mar, Región de Valparaíso
  - Hospital Clínico Regional Dr. Guillermo Grant Benavente ( Site 2604), Concepción, Región del Biobío
- China (34):
  - Anhui Provincial Hospital ( Site 3922), Hefei, Anhui
  - Peking University Third Hospital ( Site 3910), Beijing, Beijing Municipality
  - Chongqing General Hospital ( Site 3940), Chongqing, Chongqing Municipality
  - The First Affiliated Hospital Of Fujian Medical University ( Site 3916), Fuzhou, Fujian
  - The First Affiliated hospital of Xiamen University ( Site 3924), Xiamen, Fujian
  - Zhongshan Hospital Affiliated to Xiamen University ( Site 3923), Xiamen, Fujian
  - Dongguan People's Hospital ( Site 3933), Dongguan, Guangdong
  - The First Affiliated Hospital, Sun Yat-sen University ( Site 3901), Guangzhou, Guangdong
  - The Sixth Affiliated Hospital of Sun Yat-sen University ( Site 3907), Guangzhou, Guangdong
  - Huizhou Municipal Central Hospital ( Site 3915), Huizhou, Guangdong
  - Yuebei People's Hospital ( Site 3912), Shaoguan, Guangdong
  - The University of Hong Kong-Shenzhen Hospital ( Site 3930), Shenzhen, Guangdong
  - Shenzhen Hospital of Southern Medical University ( Site 3932), Shenzhen, Guangdong
  - The Second Afilliated Hospital of Hebei Medical University ( Site 3913), Shijiazhuang, Hebei
  - The Second Affiliated Hospital of Zhengzhou University ( Site 3909), Zhengzhou, Henan
  - Taihe Hospital ( Site 3944), Shiyan, Hubei
  - Renmin Hospital of Wuhan University ( Site 3921), Wuhan, Hubei
  - The Second Xiangya Hospital of Central South University-gastroenterology department ( Site 3905), Changsha, Hunan
  - Huai'an First People's Hospital ( Site 3948), Huaian, Jiangsu
  - Nanjing Drum Tower Hospital The Affiliated Hospital of Nanjing University Medical School ( Site 3937), Nanjing, Jiangsu
  - Zhongda Hospital Southeast University-Gastroenterology ( Site 3911), Nanjing, Jiangsu
  - Wuxi People's Hospital ( Site 3925), Wuxi, Jiangsu
  - Yangzhou University Affiliated Hospital ( Site 3947), Yangzhou, Jiangsu
  - Affiliated Hospital of Jiangsu University ( Site 3919), Zhenjiang, Jiangsu
  - Changzhou No.2 People's Hospital ( Site 3904), Zhenjiang, Jiangsu
  - Tangdu Hospital of Fourth Military Medical University of Chinese People's Liberation Army ( Site 3918), Xi'an, Shaanxi
  - Ruijin Hospital Shanghai Jiaotong University School of Medicine ( Site 3931), Shanghai, Shanghai Municipality
  - Huashan Hospital of Fudan University ( Site 3946), Shanghai, Shanghai Municipality
  - Shanghai East Hospital ( Site 3914), Shanghai, Shanghai Municipality
  - West China Hospital, Sichuan University ( Site 3929), Chengdu, Sichuan
  - Suining Central Hospital ( Site 3927), Suining, Sichuan
  - First Affiliated Hospital of Kunming Medical University ( Site 3928), Kunming, Yunnan
  - Sir Run Run Shaw Hospital of Zhejiang University School of Medicine-GI Medicine ( Site 3902), Hangzhou, Zhejiang
  - Taizhou Hospital of Zhejiang Province ( Site 3936), Taizhou, Zhejiang
- Colombia (6):
  - Salud SURA Industriales ( Site 2706), Medellín, Antioquia
  - Clinica Medellin S.A ( Site 2705), Medellín, Antioquia
  - Fundacion Santa Fe de Bogota ( Site 2703), Bogotá, Cundinamarca
  - IMAT S.A.S ( Site 2700), Montería, Departamento de Córdoba
  - Oncologos del Occidente ( Site 2702), Pereira, Risaralda Department
  - Fundación Valle del Lili ( Site 2704), Cali, Valle del Cauca Department
- Croatia (5):
  - Klinička bolnica Merkur ( Site 0503), Zagreb, City of Zagreb
  - Klinički bolnički centar Zagreb ( Site 0501), Zagreb, City of Zagreb
  - Poliklinika Bates ( Site 0504), Zagreb, City of Zagreb
  - Poliklinika Solmed ( Site 0502), Zagreb, City of Zagreb
  - Poliklinika Borzan ( Site 0500), Osijek, County of Osijek-Baranja
- Czechia (6):
  - KLINICKE CENTRUM Pratia Brno, Pratia Brno s.r.o. ( Site 0657), Brno, Brno-mesto
  - Vojenská Nemocnice Brno-Internal department ( Site 0655), Brno, Brno-mesto
  - Nemocnice Slany-Gastroenterologicka a Endoskopicka ambulance ( Site 0651), Slaný, Central Bohemia
  - Institut Klinicke a Experimentalni Mediciny-Klinika hepatogastroentrologie ( Site 0654), Prague, Praha 4
  - Hepato-Gastroenterologie HK ( Site 0652), Hradec Králové
  - ISCARE klinické centrum ( Site 0656), Prague
- Denmark (2):
  - Herlev and Gentofte Hospital ( Site 5300), Copenhagen, Capital Region
  - Odense Universitetshospital ( Site 5301), Odense, Region Syddanmark
- CEMDOE - Centro Médico de Diabetes, Obesidad y Especialidades ( Site 2901), Santo Domingo, Nacional, Dominican Republic
- Finland (3):
  - Tampereen yliopistollinen sairaala ( Site 5401), Tampere, Pirkanmaa
  - Pohjois-Karjalan Keskussairaala ( Site 5403), Joensuu, Pohjois-Karjala
  - Turku University Hospital ( Site 5402), Turku, Southwest Finland
- France (21):
  - Centre Hospitalier Universitaire de Nice - Hôpital l'Archet ( Site 0711), Nice, Alpes-Maritimes
  - CHU Bordeaux Haut-Leveque ( Site 0713), Pessac, Aquitaine
  - Assistance Publique Hôpitaux de Marseille - Hôpital Nord ( Site 0722), Marseille, Bouches-du-Rhone
  - Centre Hospitalier Universitaire Dijon Bourgogne - Hôpital François Mitterrand ( Site 0708), Dijon, Bourgogne-Franche-Comté
  - Centre Hospitalier Universitaire de Reims - Hôpital Robert Debré ( Site 0707), Reims, Champagne-Ardenne
  - CHU Besançon ( Site 0724), Besançon, Doubs
  - Centre Hospitalier de Valence ( Site 0725), Valence, Drome
  - C.H.U. de Nimes. Hopital Caremeau ( Site 0731), Nîmes, Gard
  - CHU Rangueil ( Site 0710), Toulouse, Haute-Garonne
  - Hopital Beaujon ( Site 0729), Clichy, Hauts-de-Seine
  - CMC Ambroise Paré Hartmann - Institut des MICI ( Site 0723), Neuilly-sur-Seine, Hauts-de-Seine
  - Clinique des Cèdres ( Site 0732), Échirolles, Isere
  - CHU SAINT ELOI ( Site 0701), Montpellier, Languedoc-Roussillon
  - Centre Hospitalier Universitaire de Nantes - L' Hopital l'hôtel-Dieu ( Site 0705), Nantes, Loire-Atlantique
  - Centre Hospitalier Régional Universitaire de Nancy - Hôpitaux de Brabois ( Site 0717), Vandœuvre-lès-Nancy, Meurthe-et-Moselle
  - Hopital Claude Huriez - CHU de Lille ( Site 0715), Lille, Nord
  - centre hospitalier lyon sud ( Site 0716), Pierre-Bénite, Rhone
  - CHU d'Amiens-Picardie - Hôpital Sud ( Site 0709), Amiens, Somme
  - Hopital Henri Mondor ( Site 0730), Créteil, Val-de-Marne
  - Hôpital Saint Antoine ( Site 0721), Paris
  - Hôpitaux Universitaires Paris Sud - Hôpital Bicêtre ( Site 0702), Le Kremlin-Bicêtre, Île-de-France Region
- Georgia (4):
  - LTD High Technology Hospital Medcenter ( Site 0802), Batumi, Adjara
  - Caucasus Medical Centre ( Site 0801), Tbilisi, Adjara
  - New Hospitals ( Site 0800), Tbilisi
  - Caraps Medline ( Site 0803), Tbilisi
- Germany (17):
  - Siloah St. Trudpert Klinikum-Zentrum für Innere Medizin ( Site 0992), Pforzheim, Baden-Wurttemberg
  - Klinikum der Universität München Großhadern ( Site 0990), München, Bavaria
  - klinikum rechts der isar der technischen universität münchen ( Site 0989), München, Bavaria
  - Universitaetsklinikum Ulm. ( Site 0994), Ulm, Bavaria
  - Medizinische Hochschule Hannover ( Site 0999), Hanover, Lower Saxony
  - Klinikum Lüneburg ( Site 0991), Lüneburg, Lower Saxony
  - Universitätsmedizin Rostock ( Site 0993), Rostock, Mecklenburg-Vorpommern
  - Evangelisches Krankenhaus Kalk gGmbH ( Site 0986), Cologne, North Rhine-Westphalia
  - Stadtische Kliniken Duisburg, Abtlg. Innere Medizin ( Site 0985), Duisburg, North Rhine-Westphalia
  - Gastroenterologische Gemeinschaftspraxis Minden ( Site 0998), Minden, North Rhine-Westphalia
  - Medizinisches Versorgungszentrum Portal 10 ( Site 0988), Münster, North Rhine-Westphalia
  - Magen Darm Zentrum Remscheid ( Site 0984), Remscheid, North Rhine-Westphalia
  - St. Marien und St. Annastift Krankenhaus ( Site 0987), Ludwighafen Am Rhein, Rhineland-Palatinate
  - Universitätsklinikum Leipzig ( Site 0997), Leipzig, Saxony
  - Universitaetsklinikum Schleswig-Holstein Campus Kiel ( Site 0995), Kiel, Schleswig-Holstein
  - Charité Campus Virchow-Klinikum ( Site 0996), Berlin
  - Universitätsklinikum Brandenburg an der Havel ( Site 0903), Brandenburg
- Greece (5):
  - Evangelismos General Hospital of Athens ( Site 1002), Athens, Attica
  - THORACIC GENERAL HOSPITAL OF ATHENS "I SOTIRIA"-3rd Dept of Internal Medicine and Laboratory, Oncol ( Site 1004), Athens, Attica
  - General Hospital of Nikaia-Piraeus "Agios Panteleimon" ( Site 1003), Nikaia Piraeus, Attica
  - Ippokrateio General Hospital of Thessaloniki ( Site 1001), Thessaloniki, Central Macedonia
  - University General Hospital of Heraklion-GASTROENTEROLOGY & HEPATOLOGY ( Site 1000), Heraklion, Crete
- Queen Mary Hospital ( Site 3300), Hksar, Hong Kong
- Hungary (10):
  - Békés Megyei Központi Kórház Dr. Réthy Pál Tagkórház-4. Belgyogyaszat Gasztroenterologia ( Site 1105), Békéscsaba, Bekescsaba
  - Heves Vármegyei Markhot Ferenc Oktatókórház és Rendelőintézet ( Site 1117), Eger, Heves County
  - Gyöngyösi Bugát Pál Kórház ( Site 1111), Gyöngyös, Heves County
  - Komarom-Esztergom Varmegyei Szent Borbala Korhaz ( Site 1115), Tatabánya, Komárom-Esztergom
  - VeszLife Magánklinika ( Site 1102), Veszprém, Veszprém megye
  - Clinexpert Kft.-Clinexpert Budapest ( Site 1108), Budapest
  - Synexus Magyarorszag Kft. (Budapest DRS) ( Site 1107), Budapest
  - Semmelweis Egyetem ( Site 1118), Budapest
  - Eszak-Pesti Centrumkorhaz-Honvedkorhaz ( Site 1100), Budapest
  - Pannónia Magánorvosi Centrum ( Site 1103), Budapest
- Beaumont Hospital, Dublin ( Site 5601), Dublin, Ireland
- Israel (9):
  - Emek Medical Center ( Site 1206), Afula
  - Barzilai Medical Center ( Site 1209), Ashkelon
  - Rambam Health Care Campus ( Site 1201), Haifa
  - Bnai Zion Medical Center ( Site 1203), Haifa
  - Edith Wolfson Medical Center ( Site 1204), Holon
  - Shaare Zedek Medical Center ( Site 1208), Jerusalem
  - Meir Medical Center. ( Site 1202), Kfar Saba
  - Rabin Medical Center ( Site 1207), Petah Tikva
  - Sheba Medical Center ( Site 1200), Ramat Gan
- Italy (15):
  - A.O.U.C. Policlinico di Bari ( Site 1306), Bari, Apulia
  - Policlinico Universitario Monserrato-SC Gastroenterologia ( Site 1313), Monserrato, Cagliari
  - Fondazione Policlinico Tor Vergata ( Site 1307), Rome, Lazio
  - Fondazione IRCCS Cà Granda Ospedale Maggiore Policlinico-Gastroenterology and Endoscopy Unit ( Site 1304), Milan, Lombardy
  - Istituto Clinico Humanitas-IBD center ( Site 1309), Rozzano, Lombardy
  - A.O.R.N. Ospedale dei Colli - Monaldi V. ( Site 1310), Naples, Napoli
  - Ospedale Mauriziano - Gastroenterology Unit ( Site 9000), Turin, Piedmont
  - Ospedale "Felice Lotti" Di Pontedera ( Site 1311), Pontedera, Pisa
  - Az. Osp. Ospedali Riuniti VILLA SOFIA-CERVELLO-U.O.S.D. Malattie Infiammatorie Croniche Intestinali ( Site 1302), Palermo, Sicily
  - Azienda Ospedaliera Universitaria Careggi-MICI ( Site 9002), Florence, Tuscany
  - Ospedale Sacro Cuore Don G. Calabria-IBD Unit ( Site 1303), Negrar, Verona
  - IRCCS Azienda Ospedaliero-Universitaria di Bologna, Policlinico di Sant'Orsola ( Site 1308), Bologna
  - Azienda Ospedaliera Universitaria Di Messina G. Martino ( Site 1314), Messina
  - Ospedale San Raffaele-Gastroenterology and Gastrointestinal Endoscopy ( Site 1300), Milan
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS -Dipartimento di Medicina Interna e Gas ( Site 1312), Roma
- Japan (55):
  - Aichi Medical University Hospital ( Site 3429), Nagakute, Aichi-ken
  - Nagoya University Hospital ( Site 3445), Nagoya, Aichi-ken
  - Nagoya City University Hospital ( Site 3446), Nagoya, Aichi-ken
  - Tokatsu Tsujinaka Hospital ( Site 3403), Abiko, Chiba
  - Tsujinaka Hospital - Kashiwanoha ( Site 3402), Kashiwa, Chiba
  - Toho University Sakura Medical Center ( Site 3413), Sakura, Chiba
  - Kurume University Hospital ( Site 3419), Kurume, Fukuoka
  - Gunma University Hospital ( Site 3432), Maebashi, Gunma
  - National Hospital Organization Fukuyama Medical Center ( Site 3442), Fukuyama, Hiroshima
  - Sapporo Tokushukai Hospital ( Site 3427), Sapporo, Hokkaido
  - Sapporo Medical University Hospital ( Site 3460), Sapporo, Hokkaido
  - Medical Corporation Sapporo IBD Clinic ( Site 3420), Sapporo, Hokkaido
  - Sapporohigashi Tokushukai Hospital ( Site 3441), Sapporo, Hokkaido
  - Hyogo Medical University Hospital ( Site 3430), Nishinomiya, Hyōgo
  - Hitachi General Hospital ( Site 3438), Hitachi, Ibaraki
  - Tsuchiura Kyodo General Hospital ( Site 3463), Tsuchiura, Ibaraki
  - Tsukuba Memorial Hospital ( Site 3461), Tsukuba, Ibaraki
  - Kanazawa University Hospital ( Site 3436), Kanazawa, Ishikawa-ken
  - Iwate Medical University Uchimaru Medical Center ( Site 3457), Morioka, Iwate
  - Gokeikai Ofuna Chuo Hospital ( Site 3412), Kamakura, Kanagawa
  - St. Marianna University Hospital ( Site 3440), Kawasaki, Kanagawa
  - Matsushima Hospital ( Site 3450), Yokohama, Kanagawa
  - Yokohama City University Medical Center ( Site 3439), Yokohama, Kanagawa
  - Mie University Hospital ( Site 3405), Tsu, Mie-ken
  - Tohoku University Hospital ( Site 3447), Sendai, Miyagi
  - University of the Ryukyus Hospital ( Site 3459), Ginowan, Okinawa
  - Kansai Medical University Hospital ( Site 3409), Hirakata, Osaka
  - Saitama Medical Center ( Site 3452), Kawagoe, Saitama
  - Hamamatsu University Hospital ( Site 3449), Hamamatsu, Shizuoka
  - Matsuda Hospital ( Site 3404), Hamamatsu, Shizuoka
  - National Hospital Organization Shizuoka Medical Center ( Site 3401), Shimizu, Shizuoka
  - Institute of Science Tokyo Hospital ( Site 3437), Bunkyō, Tokyo
  - Ginza Central Clinic ( Site 3407), Chūō, Tokyo
  - Kitasato University Kitasato Institute Hospital ( Site 3458), Minato, Tokyo
  - Toranomon Hospital ( Site 3433), Minato-ku, Tokyo
  - Kyorin University Hospital ( Site 3443), Mitaka, Tokyo
  - The Jikei University Hospital ( Site 3414), Mitato, Tokyo
  - Tokyo Medical University Hospital ( Site 3456), Shinjuku, Tokyo
  - National Center for Global Health and Medicine ( Site 3423), Shinjuku, Tokyo
  - Yamanashi Prefectural Central Hospital ( Site 3435), Kofu, Yamanashi
  - Fukuoka University Hospital ( Site 3417), Fukuoka
  - Japanese Red Cross Fukuoka Hospital ( Site 3462), Fukuoka
  - Hiroshima University Hospital ( Site 3418), Hiroshima
  - Kagoshima University Hospital ( Site 3425), Kagoshima
  - Kagoshima IBD Gastroenterology Clinic ( Site 3428), Kagoshima
  - Coloproctology Center Takano Hospital ( Site 3466), Kumamoto
  - University Hospital,Kyoto Prefectural University of Medicine ( Site 3406), Kyoto
  - National Hospital Organization Kyoto Medical Center ( Site 3411), Kyoto
  - Okayama University Hospital ( Site 3454), Okayama
  - Infusion Clinic ( Site 3408), Osaka
  - National Hospital Organization Osaka National Hospital ( Site 3453), Osaka
  - Saga University Hospital ( Site 3424), Saga
  - Tokyo Yamate Medical Center ( Site 3415), Tokyo
  - Toyama Prefectural Central Hospital ( Site 3410), Toyama
  - Yamagata University Hospital ( Site 3426), Yamagata
- Latvia (2):
  - Pauls Stradins Clinical University Hospital ( Site 5903), Riga
  - SIA M & M Centrs ( Site 5902), Ādaži, Ādaži
- Lithuania (2):
  - Hospital of Lithuanian University of Health Sciences Kauno klinikos-Gastroenterology ( Site 6000), Kaunas, Kaunas County
  - VILNIUS UNIVERSITY HOSPITAL SANTAROS KLINIKOS-Department of Clinical Trials and Pharmacology ( Site 6001), Vilnius
- Malaysia (5):
  - Hospital Sultanah Aminah ( Site 6104), Johor Bahru, Johor
  - Hospital Universiti Sains Malaysia ( Site 6103), Kubang Kerian, Kelantan
  - University Malaya Medical Centre ( Site 6101), Lembah Pantai, Kuala Lumpur
  - Sarawak General Hospital ( Site 6102), Kuching, Sarawak
  - Hospital Ampang ( Site 6106), Ampang, Selangor
- Mexico (10):
  - Morales Vargas Centro de Investigacion ( Site 3101), León, Guanajuato
  - Centro Medico Clinico Quirurgico Especializado en Investigación ( Site 3106), Tlajomulco de Zúñiga, Jalisco
  - Centro de Investigación y Gastroenterología - S.C. ( Site 3102), Mexico City, Mexico City
  - Medica Sur-Clinica de Enfermedades Digestivas y Obesidad ( Site 3104), Mexico City, Mexico City
  - JM Research SC ( Site 3109), Cuernavaca, Morelos
  - Hospital Universitario "Dr. Jose Eleuterio Gonzalez"-Gastroenterología ( Site 3100), Monterrey, Nuevo León
  - Servicios de Oncología Médica Integral, S.A de C.V. ( Site 3108), San Pedro Garza García, Nuevo León
  - Centro de Investigacion Clinica de Oaxaca ( Site 3105), Oaxaca City, Oaxaca
  - Medical Care and Research SA de CV-GASTROENTEROLOGY ( Site 3110), Mérida, Yucatán
  - Scientia Investigacion Clinica S.C. ( Site 3114), Chihuahua City
- Netherlands (8):
  - Radboudumc ( Site 1505), Nijmegen, Gelderland
  - ETZ Elisabeth ( Site 1501), Tilburg, North Brabant
  - Ziekenhuis Bernhoven ( Site 1508), Uden, North Brabant
  - Amsterdam UMC, locatie VUmc-IBD Trial Unit ( Site 1500), Amsterdam, North Holland
  - Erasmus Medisch Centrum ( Site 1504), Rotterdam, South Holland
  - Franciscus Gasthuis & Vlietland, Locatie Gasthuis ( Site 1503), Rotterdam, South Holland
  - University Medical Center Groningen ( Site 1506), Groningen
  - Universitair Medisch Centrum Utrecht ( Site 1502), Utrecht
- New Zealand (3):
  - Dunedin Hospital ( Site 3505), Dunedin, Otago
  - Hutt Valley District Health board HVDHB ( Site 3500), Lower Hutt, Wellington Region
  - Aotearoa Clinical Trials ( Site 3501), Auckland
- Peru (3):
  - Investigaciones Clínicas / Instituto de Ginecología y Reproducción ( Site 3002), Lima
  - Hospital Cayetano Heredia ( Site 3003), Lima
  - Hospital Nacional Edgardo Rebagliati Martins-Aparato Digestivo ( Site 0154), Lima
- Poland (32):
  - Pratia S.A. Pratia Poznan ( Site 1603), Poznan, Greater Poland Voivodeship
  - EMC Instytut Medyczny S.A,Prywatna Lecznica Certus Ambulatoria,Prywatna Lecznica Certus Szpital Nr1 ( Site 1605), Poznan, Greater Poland Voivodeship
  - Twoja Przychodnia Poznanskie Centrum Medyczne Sp. z o.o.,Twoja Przychodnia PCM ( Site 1632), Poznan, Greater Poland Voivodeship
  - NZOZ Centrum Medyczne KERmed ( Site 1641), Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Gastromed Sp. z o. o. ( Site 1619), Torun, Kuyavian-Pomeranian Voivodeship
  - Centrum Medyczne Plejady ( Site 1627), Krakow, Lesser Poland Voivodeship
  - FutureMeds Krakow ( Site 1628), Krakow, Lesser Poland Voivodeship
  - PROMED P. LACH R. GLOWACKI SP. J. ( Site 1636), Krakow, Lesser Poland Voivodeship
  - Allmedica ( Site 1602), Nowy Targ, Lesser Poland Voivodeship
  - Medicome Sp. z o.o ( Site 1635), Oświęcim, Lesser Poland Voivodeship
  - Amicare ( Site 1620), Jelenia Góra, Lower Silesian Voivodeship
  - Planetmed ( Site 1600), Wroclaw, Lower Silesian Voivodeship
  - Vistamed & Vertigo Sp. z o.o. ( Site 1621), Wroclaw, Lower Silesian Voivodeship
  - Melita Medical ( Site 1607), Wroclaw, Lower Silesian Voivodeship
  - Penta Hospitals Przychodnie Wrocław Wejherowska ( Site 1601), Wroclaw, Lower Silesian Voivodeship
  - Medrise Sp. z o.o. ( Site 1626), Lublin, Lublin Voivodeship
  - Uniwersytecki Szpital Kliniczny nr 4 w Lublinie, Kliniczny Oddział Gastroenterologii, Hepatologii i ( Site 1615), Lublin, Lublin Voivodeship
  - ETG Zamosc ( Site 1631), Zamość, Lublin Voivodeship
  - Centrum Zdrowia MDM ( Site 1618), Warsaw, Masovian Voivodeship
  - ETG Warszawa ( Site 1629), Warsaw, Masovian Voivodeship
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie - P-Klinika Gastroenterologii Onkologiczne ( Site 1624), Warsaw, Masovian Voivodeship
  - Vivamed Sp. z o.o. ( Site 1623), Warsaw, Masovian Voivodeship
  - WIP Warsaw IBD Point Profesor Kierkuś ( Site 1622), Warsaw, Masovian Voivodeship
  - Twoja Przychodnia Opolskie Centrum Medyczne ( Site 1633), Opole, Opole Voivodeship
  - Endoskopia Sp. z.o.o. ( Site 1637), Sopot, Pomeranian Voivodeship
  - M2M ( Site 1630), Chorzów, Silesian Voivodeship
  - H-T Centrum Medyczne Endoterapia ( Site 1610), Tychy, Silesian Voivodeship
  - Twoja Przychodnia - Szczecinskie Centrum Medyczne ( Site 1612), Szczecin, West Pomeranian Voivodeship
  - Sonomed Sp. z o. o. ( Site 1617), Szczecin, West Pomeranian Voivodeship
  - IP Clinic ( Site 1638), Lodz, Łódź Voivodeship
  - Centrum Medyczne Med-Gastr Sp. z o.o. ( Site 1616), Lodz, Łódź Voivodeship
  - AmiCare Sp. z o.o. Sp. k. ( Site 1608), Lodz, Łódź Voivodeship
- Portugal (7):
  - Unidade Local de Saúde do Alto Ave - Hospital Senhora da Oliveira ( Site 1704), Guimarães, Braga District
  - Unidade Local de Saude do Algarve - Hospital de Portimão ( Site 1700), Portimão, Faro District
  - Unidade Local de Saude da Região de Leiria - Hospital Santo André ( Site 1706), Leiria
  - Hospital da Luz Lisboa ( Site 1707), Lisbon
  - Hospital dos Lusíadas Lisboa ( Site 1701), Lisbon
  - ULSAM - Hospital de Santa Luzia ( Site 1703), Viana do Castelo
  - Unidade Local de Saude Dão-Lafões - Hospital de São Teotónio ( Site 1702), Viseu
- Romania (6):
  - MEMORIAL HEALTHCARE INTERNATIONAL S.R.L ( Site 1806), Bucharest, București
  - Fundeni Clinical Institute-Gastroenterology and Hepatology Center ( Site 1808), Bucharest, București
  - GastroMed ( Site 1809), Cluj-Napoca, Cluj
  - Spitalul Clinic Judetean Mures-Gastroenterology ( Site 1807), Târgu Mureş, Mureș County
  - ASOCIATIA ONCOHELP ( Site 1805), Timișoara, Timiș County
  - Monza Ares SRL ( Site 1804), Bucharest
- Saudi Arabia (4):
  - King Abdullah Medical City Specialist Hospital ( Site 5230), Mecca, Makkah Al Mukarramah
  - King Abdul Aziz Medical City - AlRiyadh ( Site 5210), Riyadh, Riyadh Region
  - King Saud University Medical City ( Site 5220), Riyadh, Riyadh Region
  - King Faisal Specialist Hospital and Research Center ( Site 5200), Riyadh, Riyadh Region
- Serbia (6):
  - Clinical Hospital Center Dragisa Misovic ( Site 1906), Belgrade, Beograd
  - Clinical Hospital Center Zvezdara-Gastroenterology and hepatology Department ( Site 1903), Belgrade, Beograd
  - University Medical Center "Bezanijska kosa"-Gastroenterology and hepatology ( Site 1900), Belgrade, Beograd
  - Zemun Medical Centre ( Site 1910), Zemun, Beograd
  - General Hospital "Djordje Joanovic" ( Site 1905), Zrenjanin, Srednjebanatski Okrug
  - Clinical Center Kragujevac ( Site 1904), Kragujevac, Sumadijski Okrug
- Singapore (3):
  - Singapore General Hospital ( Site 6202), Singapore, Central Singapore
  - Tan Tock Seng Hospital-Gastroenterology and Hepatology ( Site 6201), Singapore, Central Singapore
  - Changi General Hospital ( Site 6203), Singapore, South East
- Slovakia (5):
  - Fakultna nemocnica s poliklinikou F.D.Roosevelta Banska Bystrica-Gastroenterologicke oddelenie ( Site 2002), Banská Bystrica, Banská Bystrica Region
  - Cliniq s.r.o. ( Site 2001), Bratislava, Bratislava Region
  - KM Management ( Site 2000), Nitra, Nitra Region
  - GASTRO I ( Site 2004), Prešov, Presov
  - Gastro LM ( Site 2005), Prešov, Presov
- South Africa (6):
  - Wits Clinical Research ( Site 4004), Johannesburg, Gauteng
  - Wits Clinical Research-Wits Clinical Research Bara ( Site 4005), Soweto, Gauteng
  - Panorama Medical Centre ( Site 4001), Cape Town, Western Cape
  - Spoke Research ( Site 4003), Cape Town, Western Cape
  - Life Kingsbury Hospital ( Site 4000), Cape Town, Western Cape
  - Private Practice - Dr. M.N. Rajabally ( Site 4007), Plumstead, Western Cape
- South Korea (17):
  - Wonju Severance Christian Hospital-Internal Medicine ( Site 3600), Wŏnju, Kang-won-do
  - Korea University Ansan Hospital ( Site 3617), Ansan-si, Kyonggi-do
  - The Catholic University Of Korea St. Vincent's Hospital-Gastroenterology ( Site 3608), Suwon, Kyonggi-do
  - Dong-A University Hospital ( Site 3601), Busan, Pusan-Kwangyokshi
  - Inje University Haeundae Paik Hospital ( Site 3605), Haeundae-gu, Pusan-Kwangyokshi
  - Chung-Ang University Hospital ( Site 3606), Dongjak-gu, Seoul
  - Kyungpook National Univ.Hospital ( Site 3616), Daegu, Taegu-Kwangyokshi
  - Yeungnam Univeristy Medical Center ( Site 3610), Daegu, Taegu-Kwangyokshi
  - Keimyung University Dongsan Medical Center ( Site 3614), Daegu, Taegu-Kwangyokshi
  - The Catholic University of Korea, Daejeon St. Mary's Hospital ( Site 3604), Daejeon, Taejon-Kwangyokshi
  - Kyung Hee University Hospital ( Site 3611), Seoul
  - Seoul National University Hospital ( Site 3607), Seoul
  - Kangbuk Samsung Hospital-Internal Medicine ( Site 3612), Seoul
  - The Catholic University of Korea, Eunpyeong St. Mary's Hospital ( Site 3602), Seoul
  - Severance Hospital, Yonsei University Health System-Department of Internal Medicine ( Site 3603), Seoul
  - Asan Medical Center ( Site 3609), Seoul
  - Samsung Medical Center ( Site 3613), Seoul
- Spain (11):
  - Hospital Germans Trias i Pujol ( Site 2101), Badalona, Barcelona
  - HOSPITAL CLÍNIC DE BARCELONA-ICMDM - Clinical Institute of Digestive and Metabolic Diseases ( Site 2112), Barcelona, Catalonia
  - Complejo Hospitalario Universitario de Ferrol ( Site 2114), A Coruña, La Coruna
  - Hospital Universitario Puerta de Hierro ( Site 2102), Majadahonda, Madrid
  - Hospital Universitario de Torrejón ( Site 2108), Torrejón de Ardoz, Madrid
  - Hospital Universitario La Paz ( Site 2100), Madrid
  - Hospital Montecelo. Complexo Hospitalario de Pontevedra ( Site 2107), Pontevedra
  - Hospital Universitario Nuestra Senora de la Candelaria ( Site 2105), Santa Cruz de Tenerife
  - HOSPITAL CLINICO DE VALENCIA-MEDICINA DIGESTIVA ( Site 2103), Valencia
  - Hospital Universitari i Politecnic La Fe ( Site 2111), Valencia
  - Hospital Universitario Miguel Servet ( Site 2104), Zaragoza
- Sweden (3):
  - Danderyds Sjukhus ( Site 5501), Danderyd, Stockholm County
  - Karolinska Universitetssjukhuset Solna ( Site 5500), Stockholm, Stockholm County
  - Universitetssjukhuset i Linköping ( Site 5502), Linköping, Östergötland County
- Switzerland (4):
  - University Hospital Basel-Gastroenterology and Hepatology ( Site 2204), Basel, Canton of Basel-City
  - INTESTO-Gastroenterologische Praxis / Crohn-Colitis Zentrum Bern ( Site 2202), Bern, Canton of Bern
  - Cantonal Hospital St.Gallen-Klinik für Gastroenterologie / Hepatologie ( Site 2201), Sankt Gallen, Canton of St. Gallen
  - UniversitätsSpital Zürich-Gastroenterologie & Hepatologie ( Site 2200), Zurich, Canton of Zurich
- Taiwan (3):
  - National Taiwan University BioMedical Park Hospital ( Site 3702), Zhubei, Hsinchu
  - National Taiwan University Hospital-Internal Medicine ( Site 3700), Taipei
  - Chang Gung Medical Foundation-Linkou Branch ( Site 3701), Taoyuan District
- Turkey (Türkiye) (9):
  - Ege Universitesi Hastanesi ( Site 2302), Bornova, İzmir
  - Hacettepe Universitesi Tip Fakultesi Hastanesi ( Site 2300), Ankara
  - ANKARA UNIVERSITY IBNI SINA HOSPITAL-Gastroenterology ( Site 2303), Ankara
  - Ankara Bilkent Şehir Hastanesi-Gastroenterology ( Site 2301), Ankara
  - Antalya Egitim ve Arastırma Hastanesi ( Site 2304), Antalya
  - Eskisehir Osmangazi University Faculty of Medicine ( Site 2308), Eskişehir
  - Istanbul Universitesi Cerrahpasa Tip Fakultesi Hastanesi ( Site 2306), Istanbul
  - Marmara Univetsitesi Pendik Egitim ve Arastirma Hastanesi ( Site 2305), Istanbul
  - Kocaeli University Medical Faculty Hospital ( Site 2309), Kocaeli
- Ukraine (12):
  - Communal non-profit enterprise "Regional clinical hospital of Ivano-Frankivsk Regional Council" ( Site 5815), Ivano-Frankivsk, Ivano-Frankivsk Oblast
  - Medical Center of Limited ( Site 5806), Kyiv, Kyivska Oblast
  - Center of Family Medicine Plus ( Site 5803), Kyiv, Kyivska Oblast
  - Communal Non-profit Enterprise of Lviv Regional Council "Lviv Regional Clinical Hospital"-proctology ( Site 5809), Lviv, Lviv Oblast
  - Limited liability company "Medical center Health Clinic" ( Site 5807), Vinnytsia, Vinnytsia Oblast
  - Municipal Nonprofit Enterprise "Vinnytsia Regional Clinical Hospital n.a. M. I. Pyrohov of Vinnytsia ( Site 5814), Vinnytsia, Vinnytsia Oblast
  - Clinic of Scientific and Research Institute of Invalid Rehabilitation of VNMU n.a. M.I.Pyrohov ( Site 5812), Vinnytsia, Vinnytsia Oblast
  - Communal Non-Commercial Enterprise "Vinnytsia City Clinical -Clinical Therapeutic Department #1 ( Site 5811), Vinnytsia, Vinnytsia Oblast
  - Municipal Enterprise "Volyn Regional Clinical Hospital" of Volyn Regional Council ( Site 5813), Lutsk, Volyn Oblast
  - Medical Center "Universal Clinic "Oberig" of Limited Liability Company "Kapytal" ( Site 5800), Kyiv
  - Dobrobut Medical Center ( Site 5801), Kyiv
  - Medical Center of Private Enterprise "Sygma" ( Site 5808), Kyiv
- United Kingdom (10):
  - Addenbrooke's Hospital ( Site 2400), Cambridge, Cambridgeshire
  - Royal Devon & Exeter Hospital ... ( Site 2407), Exeter, Devon
  - Doncaster Royal Infirmary ( Site 2401), Doncaster, England
  - Huddersfield Royal Infirmary ( Site 2409), Huddersfield, England
  - Whipps Cross University Hospital-Clinical Research Unit ( Site 2404), London, England
  - Southampton General Hospital ( Site 2402), Southampton, Hampshire
  - University College London Hospital-Clinical Research Facility ( Site 2405), London, London, City of
  - The John Radcliffe Hospital ( Site 2406), Oxford, Oxfordshire
  - Southmead Hospital ( Site 2403), Bristol, South Gloucestershire
  - Walsall Manor Hospital ( Site 2410), West Midlands, Walsall

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26197&tenant=MT_MSD_9011